CLINICAL TRIAL: NCT06859177
Title: Remote Electrophysiological Cardiotocography (eCTG), Evaluation of Feasibility in (a Selected Group of) Complicated Pregnancies From 32 Until 37 Weeks Gestational Age in a Home@Hospital Setting: a Prospective Cohort Study
Brief Title: Feasibility of Remote eCTG Monitoring Home@Hospital in Complicated Pregnancies
Acronym: HASTA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maxima Medical Center (Other)
Collaborators: Eindhoven University of Technology (Other)
Responsible Party: Principal Investigator, Judith van Laar, Principal Investigator, Maxima Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: W24.066; PPS23-2-03529539 (Other Grant/Funding Number: PPP Allowance TKI HTSM); NL87858.015.24 (Registry Identifier: CCMO - Toetsingonline)
Record Dates: First submitted 2024-11-06; First posted 2025-03-05 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Pregnancy Related; Remote Monitoring; Feasibility
Keywords: feasibility; remote; complicated pregnancies; antenatal; Non invasive fetal electrocardiography (NI-fECG); electrophysiological cardiotocography (eCTG); high-risk pregnancies; pregnancy; maternal and fetal monitoring; monitoring; electrophysiological; non invasive; preterm pre-labor rupture of membranes (PPROM); pre-eclampsia (PE); fetal growth restriction (FGR); home monitoring; remote monitoring; second trimester; self-administered; satisfaction
MeSH Terms: conditions — Pregnancy Complications; Pre-Eclampsia; Fetal Growth Retardation; Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: Prospective single center interventional cohort study, self-administered remote electrophysiological cardiotocography (eCTG) in a home@hospital setting between 32 and 37 weeks of pregnancy, patients will complete 3 questionnaires until 4 weeks after delivery, data will be collected until 6 weeks after delivery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (1):
- Remote self-administered eCTG monitoring (using Nemo Remote®) (Experimental): Subjects will receive remote self-administered eCTG monitoring (using Nemo Remote®), daily in a Home@Hospital setting for 30-90 minutes, or at least twice weekly at the outpatient clinic.
  Interventions: Device: Remote eCTG

INTERVENTIONS:
Device: Remote eCTG — Device: Remote eCTG monitoring
  A remote self-administered electrophysiological cardiotocography (eCTG) monitoring (using Nemo Remote®), daily in a Home@Hospital setting, or at least twice weekly at the outpatient clinic, between 32 and 37 weeks of pregnancy.
  Other Names: NI-fECG

SUMMARY:
The objective of this single center, interventional cohort study is to evaluate the feasibility of remote electrophysiological cardiotocography (eCTG) monitoring in complicated pregnancies in a home@hospital setting.

The primary objective is to assess:

• The success rate of the self-administered eCTG measurement

The secondary objective is to asses:

* Maternal and perinatal outcomes
* Patients wellbeing and satisfaction.
* Healthcare professionals' (HCPs') satisfaction
* Analysis of antenatal costs

Participants will:

* Self-administer remote eCTG monitoring once daily during admission (or at least twice weekly at the outpatient clinic)
* Self-measure their blood pressure, heartrate and temperature
* Enter the measurements, symptoms and worries into an application on their telephone.
* Answer questionnaires at 3 moments during the study, assessing their wellbeing and satisfaction of the received care and self-administered remote monitoring device.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* Minimum age of 18 years old
* Pregnant patients with a gestational age between 32+0 and 36+6 weeks and days
* Singleton pregnancy
* Any indication for fetal monitoring at least twice per week (e.g.):

  * Pre-eclampsia (PE)
  * Fetal growth restriction (FGR)
  * Preterm pre-labor rupture of membranes (PPROM)
* Absence of exclusion criteria > 24 hours after admission.
* Oral and written informed consent is obtained.

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* An indication for intravenous medication
* Blood pressure >160/110 A millimeter of mercury (mmHg)
* Absent-/or reversed flow umbilical artery Doppler
* Hemolysis Elevated Liver enzymes and Low Platelets (HELLP) (Table 1)
* Obstetric intervention expected <48 hours, e.g. due to:

  * Non reassuring cardiotocography (CTG)
  * Active vaginal blood loss
  * Signs of abruption placentae
  * Meconium stained amniotic fluid
  * Signs of chorioamnionitis
* Patients admitted with a clinical diagnosis of sepsis with hypotension (i.e. septic shock).
* Insufficient knowledge of Dutch or English language
* Insufficient comprehension of instruction Nemo Remote® or patient information
* Fetal and/or maternal cardiac arrhythmias
* Contraindications to abdominal patch placement (dermatologic diseases of the abdomen precluding preparation of the abdomen with abrasive paper)
* Patients connected to an external or implanted electrical stimulator, such as Transcutaneous Electro Neuro Stimulation (TENS) and pacemaker (because of disturbance of the electrophysiological signal).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Enrollment: 60 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of successful eCTG measurements on the first day of inclusion. | On the first day of inclusion
  Count of successful* self-administered eCTG measurements on the first day of inclusion in a Home@Hospital setting, measured in numbers and percentages of total.
  1. Successful* eCTG measurement the first day at inclusion or; 2. Successful* following eCTG measurement that same day, repeated because of (reassuring but) insufficient interpretability. and no switch to conventional CTG based on interpretability was needed.
  *Successful eCTG including the following: 1. a minimum of 30 minutes eCTG registration; 2. an overall a maximum of 20% signal loss (minutes, seconds); 3. sufficient interpretability according to HCPs clinical interpretation, if not maximum extended until 90 minutes when reassuring but insufficient.

SECONDARY OUTCOMES:
Number of eCTG measurements | Inclusion up to 37 weeks of gestational age or (when earlier) up to time of delivery
  Count of eCTG measurements, measured in numbers and percentages
Number of days with eCTG measurements | Inclusion up to 37 weeks of gestational age or (when earlier) up to time of delivery
  Count of days with eCTG measurements, measured in numbers and percentages.
Number of successful eCTG measurements | Inclusion up to 37 weeks of gestational age or (when earlier) up to time of delivery
  Count of eCTG measurements assessed successful* at closure by healthcare professional, Success rate, qualified as yes or no measured in numbers and percentages of total.
  *Successful eCTG including the following: 1. a minimum of 30 minutes eCTG registration; 2. an overall a maximum of 20% signal loss (minutes, seconds); 3. sufficient interpretability according to HCPs clinical interpretation, if not maximum extended until 90 minutes when reassuring but insufficient.
  The amount of signal loss will be calculated based on the CTG. Signal loss is defined as minutes without registration of the fetal heart rate
Number of repeated eCTG measurements | Inclusion up to 37 weeks of gestational age or (when earlier) up to time of delivery
  Count of repeated eCTG measurements the same day because of reassuring but insufficient interpretability, qualified as yes or no, measured in numbers and percentages of total.
Number of switches of monitoring method from eCTG to conventional CTG monitoring, because of insufficient signal quality. | Inclusion up to 37 weeks of gestational age or (when earlier) up to time of delivery
  Count of participants in which a switch is made from eCTG to CTG monitoring because of insufficient signal quality of the eCTG measurement, qualified as yes or no, measured in numbers and percentages of total.
Switch from eCTG to conventional CTG because of maternal and/or fetal reason | Inclusion up to 37 weeks of gestational age or (when earlier) up to time of delivery
  Count of participants in which a switch is made from eCTG to CTG monitoring because of maternal and/or fetal reason, qualified as yes or no, measured in numbers and percentages of total.
Success rate of conventional CTG measurement after switch from eCTG | Inclusion up to 37 weeks of gestational age or (when earlier) up to time of delivery
  Count of successful* CTG measurements after switch from eCTG based on same criteria as in eCTG monitoring, qualified as yes or no, measured in numbers and percentages of total.
  *Successful eCTG including the following: 1. a minimum of 30 minutes eCTG registration; 2. an overall a maximum of 20% signal loss (minutes, seconds); 3. sufficient interpretability according to HCPs clinical interpretation, if not maximum extended until 90 minutes when reassuring but insufficient.
Number of eCTG measurements prematurely closed | Inclusion up to 37 weeks of gestational age or (when earlier) up to time of delivery
  Count of eCTG measurements prematurely closed by healthcare professional before complying the criteria of a successful measurement, qualified as yes of no, measured in numbers and percentages of total.
Number of participants with irritation abdominal skin | Inclusion up to 12 hours after removal last abdominal eCTG patch
  Count of patients with abdominal skin irritation, qualified as yes or no, measured in numbers and percentages of total.
Number of "unscheduled antenatal visits" | Inclusion up to 37 weeks of gestational age or (when earlier) to time of delivery
  Count of antenatal "unscheduled antenatal visits", qualified as yes or no, measured in numbers and percentages of total.
Duration of pregnancy at inclusion (days) | At inclusion
  Duration of pregnancy at inclusion, measured in days.
Maternal diagnosis at inclusion | At inclusion
  Maternal diagnosis at inclusion
Reason(s) for fetal monitoring at inclusion | At inclusion
  Reason(s) for fetal monitoring (at least 2 times a week), at the moment of inclusion (eg.
  pre-eclampsia, fetal growth restriction, preterm prelabour rupture of membranes, recurred decreased fetal movements, other reason needing monitoring at least 2 times a week)
Number of mothers admitted to the Intensive Care Unit | Inclusion up to 6 weeks post-delivery
  Count of mothers admitted to the Intensive Care Unit, qualified as yes or no, measured in numbers and percentages of total.
Number of maternal mortality | Inclusion up to 6 weeks post-delivery
  Count of maternal mortality, qualified as yes or no, measured in number and percentage in total.
Number of participants with emergency and or secondary cesarean section | Inclusion up to childbirth (up to maximum 42 weeks of gestation)
  Count of participants with emergency and or secondary cesarean section, qualified as yes or no, measured in numbers and percentages in total.
Number of participants diagnosed with abruptio placentae | Inclusion up to childbirth (up to maximum 42 weeks of gestation)
  Count of participants diagnosed with abruptio placentae, qualified as yes or no, measured in numbers and percentage of total.
Number of participants diagnosed with eclampsia | Inclusion up to 6 weeks post-delivery
  Count of participants diagnosed with eclampsia, qualified as yes or no, measured in numbers and percentages of total.
Number of participants diagnosed with HELLP syndrome | Inclusion up to 6 weeks post-delivery
  Count of participants diagnosed HELLP syndrome, qualified as yes or no, measured in numbers and percentages of total.
Number of participants diagnosed with prolapse of the umbilical cord | Inclusion up to childbirth (up to maximum 42 weeks of gestation)
  Number of participants diagnosed with prolapse of the umbilical cord, qualified as yes or no, measured in numbers and percentage of total.
Composite of maternal morbidity | Start pregnancy up to 6 weeks post-delivery
  Composite score of maternal morbidity, measured in number and percentage of one or more of the following: (eg. Emergency/secondary caesarean section, postpartum hemorrhage (bloodloss >1000ml), abruptio placentae, eclampsia, HELLP syndrome, prolapse umbilical cord, pulmonary- and/or deep venous thrombosis (combined), chorioamnionitis)
Number of perinatal mortality | Inclusion up to 7 completed days of life
  Count of fetal mortality qualified as yes or no, measured in number and percentage in total.
  General definition perinatal mortality: The number of fetal death past 22 completed weeks (154 days) of gestation plus the number of deaths among live-born children up to seven completed days of life).
Number of fetal mortality | Inclusion up to childbirth (up to maximum 42 weeks of gestation)
  Count of fetal death, qualified as yes or no, measured in numbers and percentages of total.
Number of neonatal mortality | After the seventh day but before the 28th day of life
  Count of neonatal mortality, qualified as yes or no, measured in numbers and percentages, after the seventh day up to 28 completed days of life.
Duration of pregnancy at childbirth (days) | Start pregnancy up to childbirth (up to maximum 42 weeks of gestation)
  Duration of pregnancy at childbirth, measured in days.
Number of neonates with involvement of a pediatrician | Childbirth up to 6 weeks post-delivery
  Count of participants with involvement of pediatrician, qualified as yes or no, measured in numbers and percentages of total.
Number op neonates with dysmaturity (birthweight <p3, p3-p10, <p10) | At childbirth (maximum 42 weeks of gestation)
  Count of participants with dysmaturity qualified as yes or no, measured in numbers and percentages of total.
  Based on birth weight, measured in grammes and percentiles.
  1. Below the 3th percentile; 2. From the 3th up to the 10th percentile; 3. Below 10th percentile.
Number of neonates with a congenital anomality | At childbirth
  Count of neonates with a neonatal anomality diagnosed at childbirth, qualified as yes or no, measured in numbers and percentages of total.
Number of neonates with hypoxic ischemic encephalopathy (HIE) | Childbirth up to 6 weeks post-delivery
  Count of neonates with a HIE, diagnosed at childbirth, qualified as yes or no, measured in numbers and percentages of total.
Number of neonates with Neonatal Respiratory Distress Syndrome (RDS) | Childbirth up to 6 weeks post-delivery
  Count of neonates with RDS, qualified as yes or no, measured in numbers and percentages of total.
Number of neonates with Meconium Aspiration Syndrome (MAS) | Childbirth up to 6 weeks post-delivery
  Count of neonates with MAS, qualified as yes or no, measured in numbers and percentages of total.
Number of neonates with convulsions | Childbirth up to 6 weeks post-delivery
  Count of neonates with convulsions, qualified as yes or no, measured in numbers and percentages of total.
Number of neonates with a Clinical Early Onset Sepsis (EOS) | Childbirth up to the first 72 hours, or up to 7 days after childbirth
  Number of neonates with a clinical EOS*, qualified as yes or no, measured in numbers and percentages of total.
  *Clinical early onset is defined as clinical sepsis within the first 72 hours after childbirth with > 3 days of antibiotics. Assessment from childbirth until the first 72 hours after childbirth. Or in case antibiotics later started (eg. on day 2-3) following > 3 days of antibiotics, assessment will be up to 7 days.
Number of neonates with confirmed early onset sepsis (EOS) | Childbirth up to 6 weeks post-delivery
  Count of neonates with confirmed Early Onset Sepsis (EOS) is defined as positive cultures of blood, cerebrospinal fluid, or urine from the first 72 hours after birth, qualified as yes or no, measured in numbers and percentages of total.
Number of neonates with an Apgar score at 5 minutes below 7 | 5 minutes after childbirth
  Count of neonates with an Apgar score below at 5 minutes, qualified as yes or no, measured in numbers and percentages of total.
  Apgar score (1-10) a higher score meaning a better outcome. An Apgar score of lower than 7 at 5 minutes after birth meaning a worse outcome and will be defined as asphyxia.
Number of neonates with an umbilical cord blood pH <7.05 | Directly after childbirth
  Count of neonates with an umbilical cord blood pH <7.05, meaning a severe metabolic acidosis (pH <7.05 and base deficit ≥12mmol/L), qualified as yes or no, and measured in numbers and percentages of total.
Number of neonates with neonatal asphyxia | Directly after childbirth up to 5 minutes after childbirth
  Count of neonates with neonatal asphyxia, qualified as yes or no, measured in number and percentages of total.
  Comprised one or more of the following:
  1. An Apgar score <7 at 5 minutes (Apgar score (1-10) a higher score meaning a better outcome);
  2. Umbilical cord blood pH <7.05 directly after childbirth;
  An Apgar score of lower than 7 at 5 minutes and/or an umbilical cord blood pH <7.05 after birth (combined) meaning a worse outcome and will be defined as asphyxia.
Number of neonates admitted to the Neonatal Medium Care Unit (NMCU) | Childbirth up to 6 weeks after delivery
  Count of neonates with admission to neonatal medium care unit, qualified as yes or no, measured in number and percentages of total.
Number of neonatal morbidities (composite) | Childbirth up to 6 weeks post-delivery
  Count of participants with fetal morbidity comprised one or more of the following, qualified as yes or no, and measured in number and percentages of total.
  Dysmaturity (below 3th percentile, between 3th and 10th percentile, below 10th percentile), congenital anomalies, Apgar score <7 at 5 minutes, umbilical cord blood pH <7.05, asphyxia (Apgar score <7 at 5 minutes and/or umbilical cord pH <7.05 combined)
Number of neonates with at least one neonatal diagnosis (composite) | Childbirth up to 6 weeks post-delivery
  Count of neonates with at least one neonatal diagnosis (composite), qualified as yes or no, measured in number and percentages of total.
  Complying at least one of the following: (eg. intraventricular haemorrhage (IVH), periventricular leukomalacia (PVL), bronchopulmonary dysplasia (BPD), necrotizing enterocolitis (NEC), retinopathy of prematurity (ROP), hypoxic ischemic encephalopathy, neonatal convulsions, neonatal sepsis (culture proven), needing antibiotics within the first 72 hours after birth, spontaneous intestinal perforation (SIP) necessitating surgery, surfactant treatment.
Number of neonates with the need for intubation and/or mechanical ventilation | Childbirth up to 72 hours after childbirth
  Count of neonates with the need for intubation an/or mechanical ventilation within the first 72 hours after childbirth, qualified as yes or no, measured in number and percentages of total.
Duration admission to the Neonatal Medium Care Unit (days) | Childbirth up to 6 weeks after delivery
  Duration admission to neonatal medium care unit, measured in days.
Number of neonates with an admission to the Neonatal Intensive Care Unit (NICU) | Childbirth up to 6 weeks post-delivery
  Count of neonates with the need of admission to NICU, qualified as yes or no, measured in number and percentages of total.
Duration of admission to the NICU (neonatal intensive care unit) in days. | Childbirth up to 6 weeks post-delivery
  Duration of admission to the NICU (neonatal intensive care unit), measured in days.
Assessment (twice) using a survey EuroQol including 5 dimensions and 5 levels (EQ5D-5L) to measure patient wellbeing, including visual analog pain scale (VAS) | At inclusion and at 4 weeks post-delivery
  Patient wellbeing of the given monitoring method, measured using EQ5D-5L a survey:
  This assessment tool assigns a numerical value to each response level (i.e., 1 for "no problems", 5 for "extreme problems"/"unable to") and the summing of these values across the 5 items, results in a score.
  The score is then placed on a scale, which is numbered from 0 to 100. 100 means the best health one can imagine. 0 means the worst health one can imagine.
  The questionnaire is given twice to the patient during the trial. VAS: This assessment tool assigns a score between 0 and 100 - indicating their overall health will be summarized. A higher score meaning a better health.
Assessment (once) using a surveys (D-QUEST) to measure patient satisfaction of the received monitoring method (device) | At discharge from the hospital, at 37 weeks of gestational age or (when earlier) post-delivery
  Patient satisfaction of the given monitoring method (device), measured using a survey, given once to the patient during the trial.
  Questionnaire comprises 12 items that can influence the users' satisfaction of a device and the provision process with a 5-point rating system and 2 composite items with a 5-point rating system.
  Total score range from 14 to 70, with the higher number indicating greater satisfaction.
  5-point rating: not satisfied at all (1), displeased (2), more or less satisfied (3), satisfied (4) or very satisfied (5). Personal additional information can be given in a free description space. Patients are asked to underline the 3 most important aspects of the questionnaire.
Assessment (once) using a survey (CSQ-8) to measure patient satisfaction of the overall received care | At 4 weeks post-delivery
  Client/patient satisfaction of the overall received care, measured using a survey, given once to the participants, at 4 weeks post-delivery.
  CSQ-8: comprises 8 items including scores from 1 to 4. Items 2, 4, 5, and 8 are reverse scored. Total scores range from 8 to 32, with the higher number indicating greater satisfaction.
Assessment (once) using a survey (D-Quest) to measure Healthcare professional (HCP) satisfaction of the given monitoring method. | At the moment when the last participant has delivered or has reached the gestational age of 37 weeks, assessed up to 1 month.d
  HCP satisfaction of the given monitoring method (device), measured using a survey:
  Questionnaire comprises 12 items that can influence the HCP' satisfaction of a device and the provision process with a 5-point rating system and 2 composite items with a 5-point rating system.
  Total score range from 14 to 70, with the higher number indicating greater satisfaction.
  5-point rating: not satisfied at all (1), displeased (2), more or less satisfied (3), satisfied (4) or very satisfied (5). Personal additional information can be given in a free description space. HCP are asked to underline the 3 most important aspects of the questionnaire.
  The D-Quest survey is based on a validated patient questionnaire and suitable for HCPs after minimal adjustments. HCP will receive the survey once, at the moment when the last participant has delivered or has reached the gestational age of 37 weeks.
Antenatal costs as a business case model | Inclusion up to moment of start delivery (antenatal period), assessed up to maximum 42 weeks of gestation.
  To assess the costs (euro) of remote home monitoring versus in-hospital monitoring, patient journeys will be followed and costs calculated (N,n, Euro) as if they were at home using remote eCTG compared to in- hospital standard care using conventional CTG. (eg. eCTG, CTG, admission day, visits, emergency ambulance rides)
  The patient journey will not depend on participation in the HASTA study but is part of the standard care and HCP decision.
  Total of costs: mean and median (euro) and the percentage (%) of patients with at least one registered activity (% treated). In addition, a sub-analysis will be presented of participants needing hospitalization and of participants monitoring at the outpatient clinic at inclusion.

OTHER OUTCOMES:
Number of participants with analgesia for pain reduction: epidural or/and remifentanil | During delivery
  Count of participants with analgesia for pain reduction during delivery, qualified as yes or no, measured in numbers and percentages of total.
Number of participants with perineal laceration | Directly after childbirth
  Count of participants with perineal laceration (grade 1, 2, 3a, 3b, 3c, 4), qualified as yes or no, measured in numbers and percentage of total.
Number of participants with an episiotomy | Directly after childbirth
  Count of participants with an episiotomy, qualified as yes or no, measured in numbers and percentages of total.
Number of mothers with an obstetric haemorrhage | Childbirth up to 24 hours after childbirth
  Count of mothers with an obstetric haemorrhage, qualified as yes or no, measured in numbers and percentages of total. Obstetric haemorrhage > 1000 millilitres within 24 hours after giving birth
Number of mothers with a thromboembolic event | Inclusion up to 6 weeks post-delivery
  Count of mothers with a thromboembolic event, qualified as yes or no, measured in numbers and percentages of total. (pulmonary- and/or deep venous thrombosis (combined))
Number of mothers with an uterine rupture | Childbirth up to 6 weeks post-delivery
  Count of mothers with an uterine rupture, qualified as yes or no, and measured in numbers and percentages of total.
Number of mothers with a suspected or confirmed postpartum infection requiring antibiotics | Childbirth up to 6 weeks post-delivery
  Count of mothers with a suspected or confirmed postpartum infection requiring antibiotics, qualified as yes or no, measured in numbers and percentages in total. (eg. post-delivery infection requiring antibiotics: urinary tract infection, chorioamnionitis, endometritis, infection following CS, pneumonia, mastitis).
Number of mothers with a postpartum anemia due to postpartum haemorrhage with requires red cell transfusion | Childbirth up to 6 weeks post-delivery
  Count of mothers with a postpartum anemia due to postpartum haemorrhage with requires red cell transfusion, qualified as yes or no, measured in numbers and percentages in total.

CONTACTS AND LOCATIONS:
Overall Officials: Judith O.E.H. van Laar, MD, PhD, Principal Investigator — Máxima Medical Center, Technical University of Eindhoven
Locations (1):
- Maxima Medical Center, Veldhoven, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, anonymous data, Informed Consent Form, general assessment and registration formulary
Supporting Information: Study Protocol, ICF
Time Frame: When requested and after assessment, the anonymous data - presented in this study - will be shared with researchers conducting pregnancy related studies after publication of the study results in a medical journal .
  Study protocol will be submitted for publication and will be available once published.
  All data will be stored at Maxima Medical Center (MMC) in Veldhoven, in The Netherlands, for at least 15 years after completion of the study, this is a legal obligation.
Access Criteria: Anonymous data: researchers conducting pregnancy related studies. Informed Consent Form: researchers conducting pregnancy related studies. Protocol: when admitted for publication, open access.
URL: http://www.toetsingonline.nl/to/ccmo_search.nsf/fABRpop?readform&unids=5E9DC57EAB3DCF44C1258BCD0005C711

REFERENCES:
- [Derived] van Weelden S, Monen L, van der Hout-van der Jagt MB, van Laar JOEH. Remote electrophysiological cardiotocography (eCTG), evaluation of feasibility in complicated pregnancies from 32 until 37 weeks gestational age in a home@hospital setting (HASTA): A prospective cohort study protocol. PLoS One. 2026 Feb 3;21(2):e0341554. doi: 10.1371/journal.pone.0341554. eCollection 2026. PMID 41632811
- See also: Central Committee on Human Research — https://www.toetsingonline.nl/to/ccmo_search.nsf/fABRpop?readform&unids=5E9DC57EAB3DCF44C1258BCD0005C711